CLINICAL TRIAL: NCT03675464
Title: Longitudinal Observational Study of Human Adipose Tissue (LOSHAT)
Brief Title: Study of Human Adipose Tissue (LOSHAT)
Acronym: LOSHAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Peter Arner, Professor, Karolinska University Hospital
Other Study IDs: 2018/809-31
Record Dates: First submitted 2018-08-23; First posted 2018-09-18 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Weight Change, Body; Weight Loss; Weight Gain; Lipolysis; Adipose Tissue; Human; Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Body Weight Changes; Weight Loss; Weight Gain; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will study the influence of initial fat cell size/number and adipose function (in particular lipolysis) on weight development over very long time periods (years). By comparing investigations of fat biopsies or blood samples obtained at baseline, the investigators will determine the association between adipose morphology/function and changes in weight or development of metabolic complications (e.g. metabolic syndrome, glucose intolerance, type 2 diabetes, dyslipidemia and hypertension).

DETAILED DESCRIPTION:
The investigators will ask all subjects that have previously been examined at the investigators laboratory (from 1992 and forward) in studies of adipose tissue function if they are interested to participate in a new study.

Previously obtained results from examinations of adipose tissue, anthropometric measurements and blood samples will be used as baseline. In addition, saved blood samples and samples from old fat biopsies can be re-investigated in some cases.

The new investigation includes a questionnaire that the subjects can answer by mail or email. In addition, anthropometric measurements and blood pressure determination will be performed at a primary health care center and blood samples will be collected for analysis of fasting glucose, HbA1C and lipids.

Information regarding all previously investigated subjects will also be collected from several Swedish national patient registries such as the Patient Register, Prescribed Drug register and Cause-of Death register.

ELIGIBILITY:
Inclusion Criteria:

* Previously participated in examinations at the investigators laboratory and donated adipose tissue.
* Previously participated in examinations at the investigators laboratory and donated blood samples that can be used to estimate lipolysis with a formula.

Exclusion Criteria:

* Decline to participate after invitation.
* Severe Psychiatric disease.
* Type 1 Diabetes
* Participants that have undergone bariatric surgery will be exluded in the primary analysis but will be analyzed separately in a secondary analysis for all above mentioned outcomes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women previously examined at our laboratory
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Body mass index | 2018 to 2022
  Body weight (in kilogram) will be assessed with a regular scale. Height will be measured with a tape measure (in centimeters). Body mass index (BMI) will be calculated with the formula weight (kg) divided by height^2 (in meter). Changes in BMI from baseline values will be analysed.
Fasting glucose | 2018 to 2022
  Fasting plasma glucose will be assessed and divided into normal glucose (glucose < 6.1 mmol/L), impaired fasting glucose (glucose 6.1-6.9 mmol/L) or type 2 diabetes (glucose > 6.9 mmol/L).
Number of participants with metabolic syndrome | 2018 to 2022
  Metabolic syndrome is defined according to International Diabetes Federation, Waist circumference ≥102 cm for men or ≥88 cm for women. In addition to this 2 of the following; Raised triglycerides: > 150 mg/dL (1.7 mmol/L), or specific treatment for this lipid abnormality; Reduced HDL cholesterol: < 40 mg/dL (1.03 mmol/L) in males, < 50 mg/dL (1.29 mmol/L) in females, or specific treatment for this lipid abnormality; Raised blood pressure (BP): systolic BP > 130 or diastolic BP >85 mm Hg, or treatment of previously diagnosed hypertension; Raised fasting plasma glucose (FPG): >100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes. Scores are 0-5. ≥ 3 is defined as metabolic syndrome.
Number of participants with type 2 Diabetes | 2018 to 2022
  Based on a diagnosis in the Swedish National Patient Register, or prescribed drugs for Type 2 diabetes in the Swedish National Prescribed Drug Register or direct information from the subject.
Number of participants with dyslipidemia | 2018 to 2022
  Based on a diagnosis in the Swedish National Patient Register, or prescribed drugs for dyslipidemia in the Swedish National Prescribed Drug Register, or direct information from the subject.
Number of participants with Hypertension | 2018 to 2022
  Based on a diagnosis in the Swedish National Patient Register, or prescribed drugs for hypertension in the Swedish National Prescribed Drug Register, or direct information from the subject.

SECONDARY OUTCOMES:
Genetic variations linked to lipolysis | 2018 to 2022
  Genome-wide association study (GWAS) with focus on genes related to lipolysis and analysis of single nucleotide polymorphisms (SNPs). Samples from baseline examination will be used in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Arner, MD, PhD, Principal Investigator — Karolinska University Hospital; Daniel P Andersson, MD, PhD, Study Director — Karolinska University Hospital; Mikael Rydén, Md, PhD, Study Chair — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden